CLINICAL TRIAL: NCT07042568
Title: The Effect of Education Given to Women Diagnosed With Breast Cancer to Prevent Oral Mucositis on Quality of Life
Brief Title: The Effect of Education Given on Preventing Mouth Ulcers in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, YAREN ÖZBEK, Research Assistant, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TÜTF-GOBAEK 2022/382
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Chemotherapy
Keywords: Education; Breast cancer; Chemotherapy; Oral mucositis; Quality of life; Nursing
MeSH Terms: conditions — Breast Neoplasms; Stomatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Education + Telephone consultation) (Experimental)
  Interventions: Behavioral: Nursing education aimed at preventing oral mucositis
- Control group (No Intervention): They continued to receive routine nursing care.

INTERVENTIONS:
Behavioral: Nursing education aimed at preventing oral mucositis — The intervention group was trained on the use of the Oral Mucositis Prevention Patient Education Handbook, which was prepared by the researchers based on literature information and expert opinions. Participants in the intervention group received telephone consultations on days 7 and 14. The control group continued to receive routine nursing care. The second interview was completed on day 21, when both the intervention and control group patients returned for their next treatment cycle, using the WHO Oral Toxicity Criteria, ADR, and EORTC QLQ-C30 Version 3.0 Quality of Life Scale.
  Arms: Intervention (Education + Telephone consultation)

SUMMARY:
This study aims to evaluate the effect of nursing education provided to women diagnosed with breast cancer undergoing chemotherapy on their quality of life and the severity of oral mucositis (mouth sores).

The main questions this study aims to answer are:

1. Does nursing education aimed at preventing oral mucositis in women diagnosed with breast cancer have an effect on quality of life?
2. Does nursing education aimed at preventing oral mucositis in women diagnosed with breast cancer have an effect on the severity of oral mucositis? The researchers will evaluate the effect of nursing education on quality of life and oral mucositis severity by randomly assigning one group to receive education and the other group to not receive education.

Participants:

When they come to receive their chemotherapy treatment (on the first day of the evaluation), the researcher will fill out a scale measuring quality of life and scales checking the condition of the oral mucosa. Participants in the education group will receive education from the researchers using an education booklet prepared by the researchers, and the booklet will remain with the participants. On days 7 and 14, the researcher will provide telephone consultation. On the 21st day, when the final evaluation will be conducted, data will be collected from participants through the scales.

DETAILED DESCRIPTION:
This study is a two-armed, single-blind, randomised controlled trial (RCT). Participants were selected from an oncology hospital affiliated with a university hospital in western Turkey between February and August 2023. Women who met the following criteria were included in the study: Women diagnosed with breast cancer who were undergoing chemotherapy, aged 18 years or older, voluntarily participating in the study, capable of communicating in Turkish, and able to read and write, with at least three weeks of chemotherapy treatment remaining.

Patients who met the following criteria were excluded from the study: having a known psychiatric disorder that could interfere with the intervention and data collection process, receiving chemoradiotherapy, or having cognitive, perceptual, or communication problems that could affect their ability to understand the training provided.

To determine the sample size, a pre-power analysis was performed using the G-Power 3.1.9.7 programme. For this analysis, the initial measurement total mean EORTC QLQ-C30 quality of life scale scores of the intervention and control groups in the study by Yüce and Yurtsever [24] were used. According to the analysis results, with an effect size of 0.65, a significance level of p<0.05 in each group, a 95% confidence interval, and 80% test power, a minimum of 78 participants (39 participants each for the intervention and control groups) was determined. A total of 91 patients were reached during the specified dates, but 6 patients did not wish to continue the study and were therefore not included in the analysis. The study was completed with a total of 85 participants, including 43 in the intervention group and 42 in the control group.

After obtaining the necessary ethical committee and institutional approvals for this study, it was conducted through face-to-face interviews in a suitable room in the outpatient chemotherapy unit on the first day and the 21st day of chemotherapy for female patients diagnosed with breast cancer who met the inclusion criteria. On the first day of the interview, all participants were informed about the purpose and method of the study, and it was emphasised that participation in the study was entirely voluntary. Written informed consent was obtained through an informed consent form.

Taking into account the order of the randomisation table, one participant was included in the study each day, and on the first day of the interview, the researchers administered the Patient Information Form, the World Health Organisation (WHO) Oral Toxicity Criteria, the Oral Assessment Guide (OAG), European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) Version 3.0 Quality of Life Scale, Eastern Cooperative Oncology Group (ECOG) Performance Scale. In addition, the intervention group was trained on the use of the Oral Mucositis Prevention Patient Education Handbook, which was prepared by the researchers based on literature information and expert opinions. Participants in the intervention group received telephone consultations on days 7 and 14. The control group continued to receive routine nursing care. The second interview was completed on day 21, when both the intervention and control group patients returned for their next treatment cycle, using the WHO Oral Toxicity Criteria, ADR, and EORTC QLQ-C30 Version 3.0 Quality of Life Scale.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer and undergoing chemotherapy,
* Aged 18 or older,
* Volunteering to participate in the study,
* Able to communicate, read and write in Turkish,
* With at least 3 weeks of chemotherapy treatment remaining

Exclusion Criteria:

* Having a known psychiatric illness that could interfere with the intervention and data collection process,
* Receiving chemo-radiotherapy,
* Having cognitive, perceptual, or communication issues that may affect their ability to understand the provided education.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Comparison of general health, functional and symptom-related quality of life (QLQ-C30), WHO oral toxicity criteria and ADR measurement scores within and between the intervention and control groups | First day and 21st day
  The European Organisation for Research and Treatment of Cancer QLQ-C30 Version 3.0 Quality of Life Scale consists of a total of 30 questions divided into three subscales: general well-being, functional scale, and symptom scale.
  In this scale developed by the WHO, stage 0 represents normal oral mucosa, while stage 4 represents the highest severity of oral mucositis.
  The Oral Assessment Guide (OAG) covers eight areas: voice, swallowing, tongue, lips, oral mucosa, saliva, gums, and teeth/dentures. When calculating the final total oral mucosa score, the scores obtained from these eight areas are added together. The lowest score is 8, and the highest score is 24. An increase in the score indicates an increase in the severity of oral mucositis, while a decrease indicates a decrease in the severity of oral mucositis.

CONTACTS AND LOCATIONS:
Locations (1):
- Balkan Oncology Hospital affiliated with Trakya University Hospital, Trakya University, Republic of Turkey, Edirne, Turkey (Türkiye)